CLINICAL TRIAL: NCT03235440
Title: Examination of the Acceptance and Feasibility of Implementing the American Diabetes Association's Camp Power Up Program on Changes in Body Weight and Quality of Life Measures in Children
Brief Title: Feasibility of the Camp Power Up Program on Children's Body Weight and Quality of Life
Acronym: CampPowerUp
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: American Diabetes Association (Other); Louisiana State University, Baton Rouge (Other); American Council on Exercise (Other)
Responsible Party: Principal Investigator, Amanda Staiano, Assistant Professor - Research, Pennington Biomedical Research Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PBRC 2017-014
Record Dates: First submitted 2017-07-21; First posted 2017-08-01 (Actual); Results first posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-11

CONDITIONS: Obesity, Childhood; Weight Change, Body; Quality of Life
MeSH Terms: conditions — Pediatric Obesity; Body Weight Changes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Kids N Fitness (Experimental): Participants will engage in a one-week weight-management summer camp consisting of different activities related to moderate-vigorous physical activity (MVPA) and healthy eating. MVPA will consist of modifiable games and activities using a variety of equipment familiar to children of this age, such as balls, hula-hoops, Frisbees, etc., in both competitive and cooperative formats that keep participants moving at all times, and emphasize a feeling of play as opposed to a feeling of exercise. Healthy eating activities are composed of varying classroom-style learning and practical application of knowledge to topics such as recommendations from the MyPlate.gov website, the different types of food groups, and caloric intake and portion sizes, among other various topics.
  Interventions: Behavioral: Kids N Fitness Program

INTERVENTIONS:
Behavioral: Kids N Fitness Program — Participants will engage in a one-week weight-management summer camp consisting of different activities related to moderate-vigorous physical activity (MVPA) and healthy eating. MVPA will consist of modifiable games and activities using a variety of equipment familiar to children of this age, such as balls, hula-hoops, Frisbees, etc., in both competitive and cooperative formats that keep participants moving at all times, and emphasize a feeling of play as opposed to a feeling of exercise. Healthy eating activities are composed of varying classroom-style learning and practical application of knowledge to topics such as recommendations from the MyPlate.gov website, the different types of food groups, and caloric intake and portion sizes, among other various topics.
  Other Names: Kids N Fitness (KNF) Program

SUMMARY:
This study will evaluate the effects of a one week weight management summer camp on children's weight, quality of life, mood and feelings, self-esteem, weight management efficacy, enjoyment of physical activity, and body image.

DETAILED DESCRIPTION:
Obesity affects 17% of children and adolescents in the U.S. Children are entrenched in an obesogenic environment, often with little support in the home, school, or medical environment to make healthy choices. Obesity is increasingly common in underserved communities that lack access and resources for physical activity and healthy eating. Louisiana is a prime example of the need for effective obesity treatment, ranking 1st nationally for adult obesity and 4th for adolescent obesity with the highest obesity prevalence among African American adolescents. We urgently need evidence-based programs to help children and families change lifestyle behaviors, achieve clinically significant weight loss, and thereby reduce the prevalence of pediatric obesity.

The U.S. Preventive Services Task Force identifies behavioral treatment including dietary, physical activity, and behavioral counseling components as a viable option for pediatric obesity treatment, yet a key challenge is how to implement these programs to maximize access and participation. Summer (between school years) represents an opportunity for intensive intervention to change health behaviors and help children to lose weight. During the summer months, children gain weight at a more rapid pace and spend more time engaged in sedentary behavior compared to the school year.

The American Diabetes Association launched Camp Power Up as a summer week-long day camp for youth who are obese and/or at high risk for developing type 2 diabetes. The camp will focus on wellness education, nutrition, physical activity, and obesity prevention. The purpose of the proposed study is to examine effects of Camp Power Up on children's weight status and their psycho-social health.

ELIGIBILITY:
Inclusion Criteria:

* Aged 6 to 14 years
* Enrolled in the American Diabetes Association (ADA) Camp Power Up

Exclusion Criteria:

-

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 27 (Actual)
Dates: Start 2017-06-19 (Actual); Primary Completion 2018-06-15 (Actual); Study Completion 2018-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amanda E Staiano, Ph.D., Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Kids N Fitness: Participants will engage in a one-week weight-management summer camp consisting of different activities related to moderate-vigorous physical activity (MVPA) & healthy eating. MVPA will consist of modifiable games & activities using a variety of equipment familiar to children of this age, such as balls, hula-hoops, etc., in both competitive & cooperative formats that keep participants moving at all times, & emphasize a feeling of play as opposed to a feeling of exercise. Healthy eating activities are composed of varying classroom-style learning & practical application of knowledge to topics such as recommendations from the MyPlate.gov website, the different types of food groups, & caloric intake and portion sizes, among other various topics.
Period: Overall Study
Arm/Group | Kids N Fitness
Started | 27
Completed | 24
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Kids N Fitness
Number analyzed (Participants) | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 27
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 13
  More than one race | 5
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Body Weight
Description: Weight measurement (kg) using a standard scale following the Pennington Biomedical Standard Operating Procedure for weight measurements.
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Kids N Fitness
Number analyzed (Participants) | 24
kg | .3 (.5)

2. Secondary Outcome: Impact of Weight on Quality of Life (IWQOL): IWQOL-Kids
Description: The Impact of Weight on Quality of Life-Kids (IWQOL-Kids) is a validated self-report measure designed to assess weight-related quality of life in adolescents aged 11-19. It includes four subscales-physical comfort, body esteem, social life, and family relations-along with a total score, all of which show strong psychometric properties. Response options range from always true (1) to never true (5). Total scores range from 0-135, where higher scores represent better health-related quality of life.
Time Frame: 5 Days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Kids N Fitness
Number analyzed (Participants) | 11
score on a scale
  Pre (day 1) | 123.7 (12.2)
  Post (day 5) | 128.6 (13.7)

3. Secondary Outcome: Pediatric Quality of Life Inventory - PedsQL
Description: A method of measuring health-related quality of life (HRQOL) in children between ages 2-18 years that are either healthy or have health conditions. They are flexible in use and are multidimensional, covering physical, emotional, social, and school functioning. The measure consists of four core scales (physical, emotional, social, and school), two broad domain scores (physical and psychosocial functioning), and a total score. The PedsQL uses a 5-point Likert scale for responses (Never a problem, Almost never a problem, Sometimes a problem, Often a problem, and Almost always a problem). Scales are standardized, and scores range from 0 to 100, with higher scores representing better quality of life.
Time Frame: First day and final day of camp (day 1 and day 5)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Kids N Fitness
Number analyzed (Participants) | 11
score on a scale
  Pre (day 1) | 80.5 (16.9)
  Post (day 5) | 84.3 (13.7)

4. Secondary Outcome: Weight Efficacy Lifestyle Questionnaire (WEL)
Description: A self-report measure designed to assess an individual's confidence in their ability to control eating behavior in various situations, such as during negative emotions, social pressures, or availability of food. Subjects were asked to rate their confidence on being able to resist the urge to eat using a Likert scale ranging from 0 (not confident) to 9 (very confident); the total score for the WEL is the sum of all 20 items, giving a range of 0 to 180. Higher total scores (closer to the maximum of 180) and higher subscale scores reflect a greater sense of confidence in one's ability to resist eating in challenging situations. Lower total scores (closer to the minimum of 0) and lower subscale scores indicate less confidence in resisting eating in challenging situations.
Time Frame: First day and final day of camp (day 1 and day 5)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Kids N Fitness
Number analyzed (Participants) | 11
score on a scale
  Pre (day 1) | 52.0 (21.2)
  Post (day 5) | 48.3 (24.9)

5. Secondary Outcome: Physical Activity Enjoyment Scale (PACES)
Description: A self-report tool used to measure an individual's enjoyment of physical activity. It assesses the positive feelings and overall satisfaction associated with engaging in exercise. Respondents are asked to rate "how you feel at the moment about the physical activity you have been doing" using a 7-point bipolar rating scale (1-7) on 18 items. Eleven items are reverse scored where the score values are flipped (i.e., 1=7, 2=6, …). Higher total PACES scores demonstrate greater levels of enjoyment. The lowest possible score is 18 while the highest is 126.
Time Frame: First day and final day of camp (day 1 and day 5)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Kids N Fitness
Number analyzed (Participants) | 11
score on a scale
  Pre (day 1) | 47.8 (13.7)
  Post (day 5) | 52.6 (7.4)

6. Secondary Outcome: Body Image Assessment of Children (BIA-C):
Description: A tool used to evaluate children's perceptions of their body size and shape. It helps identify body image concerns by comparing their self-perceived body figure with a body figure that represents their ideal figure. The scale ranges from 1 to 9, each number representing a body size. A body dysphoria score is derived from the difference between the current body state and ideal body state (CBS - IBS) the participant chooses. Positive scores (where the current size is larger than the ideal) may indicate a desire to be thinner, while negative scores (where the current size is smaller than the ideal) may indicate a desire to be larger. Scores range from -5 to +5. Negative scores indicate a preference for a larger body size than the perceived size. Positive scores indicate a preference for a smaller body size than the perceived size. Scale numbers were combined based on the average total score.
Time Frame: First day and final day of camp (day 1 and day 5)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Kids N Fitness
Number analyzed (Participants) | 11
score on a scale
  Pre (day 1) | 2.3 (1.8)
  Post (day 5) | 1.9 (1.9)

ADVERSE EVENTS:
Time Frame: 1 week
Arm/Group | Kids N Fitness
All-Cause Mortality (participants affected / at risk) | 0/27
Serious Adverse Events (participants affected / at risk) | 0/27
Other Adverse Events (participants affected / at risk) | 0/27

LIMITATIONS AND CAVEATS:
Without being limited to one week in favor of an entire summer, the results could show significant improvements in multiple categories, including physical activity and weight status. Camp Power aimed to improve psychosocial health of the children as well. Only one week showed marginal changes in health-related quality of life.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-09-01): https://cdn.clinicaltrials.gov/large-docs/40/NCT03235440/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-01): https://cdn.clinicaltrials.gov/large-docs/40/NCT03235440/SAP_001.pdf